CLINICAL TRIAL: NCT03212391
Title: Effect of Diet and Physical Exercise, With or Without Nordic Walking, on Weight Loss, Physical Performance and Cardiovascular Risk Factors in Elderly Overweight and Obese Subjects.
Brief Title: WAVE Study- Walking and Aging in VErona Study
Acronym: WAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 739CESC
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Abdominal Obesity; Metabolic Syndrome; Disability Physical; Sarcopenic Obesity; Hypertension; Overweight and Obesity; Cardiovascular Risk Factor
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome; Hypertension; Overweight; Obesity | interventions — Diet; Walking; Nordic Walking

STUDY DESIGN:
Intervention Model Description: Monocentric unblinded two parallel-group randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet+Walking (Experimental): 52 weeks of Diet+26 weeks supervised Walking 3 times per week, followed by 26 weeks of unsupervised Walking
  Interventions: Behavioral: Diet; Behavioral: Walking
- Diet+Nordic Walking (Experimental): 52 weeks of Diet+26 weeks supervised Nordic Walking 3 times per week, followed by 26 weeks of unsupervised Nordic Walking
  Interventions: Behavioral: Diet; Behavioral: Nordic Walking

INTERVENTIONS:
Behavioral: Diet — 52 weeks of Diet supervised by a dietician
Behavioral: Walking — 26 weeks supervised Walking 3 times per week, followed by 26 weeks of unsupervised Walking
  Arms: Diet+Walking
Behavioral: Nordic Walking — 26 weeks supervised Nordic Walking 3 times per week, followed by 26 weeks of unsupervised Nordic Walking
  Arms: Diet+Nordic Walking

SUMMARY:
Monocentric unblinded two parallel-group randomized controlled trial to evaluate the effect of diet with or without Nordic Walking on weight loss, physical performance and cardiovascular risk factors in overweight and obese population

DETAILED DESCRIPTION:
To examine the impact of a 48-week of diet +/- Nordic Walking program on physical performance, muscle function, cardiovascular risk factors and arterial stiffness in community-dwelling overweight and obese elderly men and women.

ELIGIBILITY:
Inclusion Criteria:

* 60-90 years

  * Males and females

    . BMI > 27 kg/m2
  * living in Verona (Italy)
  * stable weight in the 3 months
  * not involved in physical exercise programs
  * informed consent sign

Exclusion Criteria:

* cardiovascular disease (unstable angina, recent myocardial infarction, cardiac arrhythmias, heart failure, valvular heart disease, aortic aneurysm, recent intracerebral or subdural hemorrhage, not controlled hypertension)
* musculoskeletal disease (symptomatic discal hernia, symptomatic arthrosis, acute articular, tendon or ligament lesions, hip prothesis).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-09-19 (Actual); Primary Completion 2018-01-20 (Estimated); Study Completion 2018-07-20 (Estimated)

PRIMARY OUTCOMES:
VO2 max | 12 months
  maximal oxygen consumption

SECONDARY OUTCOMES:
VO2 max changes | 3, 6, 9 and 12 months
  maximal oxygen consumption
PWV | 3, 6, 9 and 12 months
  pulse wave velocity
muscle strength | 3, 6, 9 and 12 months
fat mass | 3, 6, 9 and 12 months
muscle mass | 3, 6, 9 and 12 months
SF 36 | 6 and 12 months
  quality of life
GDS | 6 and 12 months
  geriatric depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Zamboni, Study Director — AOUI Verona
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muollo V, Rossi AP, Milanese C, Zamboni M, Rosa R, Schena F, Pellegrini B. Prolonged unsupervised Nordic walking and walking exercise following six months of supervision in adults with overweight and obesity: A randomised clinical trial. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1247-1256. doi: 10.1016/j.numecd.2020.12.012. Epub 2020 Dec 17. PMID 33549445